CLINICAL TRIAL: NCT00453791
Title: A Randomised, Single and Repeat Dose, Double-blind, Placebo Controlled Study to Assess the Safety and Tolerability of GW805858 in Healthy Volunteers and Mild Asthmatics
Brief Title: The Safety and Tolerability of GW805858 in Healthy Volunteers and Mild Asthmatics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: SF2105450
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: GW805858; MDI; asthma; surfactant
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Subjects receiving treatment sequence 1: Part 1 (Experimental): Eligible subjects will receive placebo followed by GW805858 with a starting dose of 150 micrograms administered using Metered Dose Inhaler (MDI).
  Interventions: Drug: GW805858; Drug: Placebo
- Subjects receiving treatment sequence 2: Part 1 (Experimental): Eligible subjects will receive GW805858 with a starting dose of 150 micrograms followed by placebo administered using MDI.
  Interventions: Drug: GW805858; Drug: Placebo
- Subjects receiving treatment sequence 1: Part 2 (Experimental): Eligible subjects will receive placebo followed by GW805858 with a starting dose of 150 micrograms administered using MDI.
  Interventions: Drug: GW805858; Drug: Placebo
- Subjects receiving treatment sequence 2: Part 2 (Experimental): Eligible subjects will receive GW805858 with a starting dose of 150 micrograms followed by placebo administered using MDI.
  Interventions: Drug: GW805858; Drug: Placebo
- Subjects receiving GW805858: Part 3 (Experimental): Eligible subjects will receive GW805858 1200 micrograms twice daily administered using MDI.
  Interventions: Drug: GW805858
- Subjects receiving placebo: Part 3 (Experimental): Eligible subjects will receive placebo administered using MDI.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW805858 — GW805858 MDI will be given with dose of 150 micrograms per metered actuation and 120 actuations per inhaler. GW805858 MDI comprises a solution of GW805858 in a liquefied hydrofluoroalkane propellant (1,1,1,2-tetrafluoroethane) which is contained in an aluminium alloy can, internally coated with a specified fluoropolymer, fitted with a metering valve.
  Arms: Subjects receiving GW805858: Part 3; Subjects receiving treatment sequence 1: Part 1; Subjects receiving treatment sequence 1: Part 2; Subjects receiving treatment sequence 2: Part 1; Subjects receiving treatment sequence 2: Part 2
Drug: Placebo — Placebo MDI will be given to the subjects.
  Arms: Subjects receiving placebo: Part 3; Subjects receiving treatment sequence 1: Part 1; Subjects receiving treatment sequence 1: Part 2; Subjects receiving treatment sequence 2: Part 1; Subjects receiving treatment sequence 2: Part 2

SUMMARY:
This study will be the First Time in Human Study (FTIH) aiming to assess the safety and tolerability of GW805858 for both single and repeat dose. The study also aims to assess safety and tolerability in mild asthmatic subjects as well as healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-child bearing potential, aged between 18 and 60 years of age inclusive.
* Body weight = 50 kg (110 lbs) for men and = 45 kg for women and Body Mass Index (BMI) within the range 19.0-30.0 kg/m2 inclusive.
* The subject is a current non-smoker who has not used any tobacco products in the last year.
* A signed and dated written informed consent is obtained for the subject.
* The subject is able to understand and comply with protocol requirements and timetables, instructions and protocol-stated restrictions.
* If asthmatic, the subject must be a clinically stable asthmatic.

Exclusion Criteria:

* The subject has a history of allergy to ingredients within the inhaler.
* The subject has received an investigational drug or participated in any other research trial within 30 days, prior to the first dose of current study medication.
* The subject has used prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days prior to the first dose of study medication.
* The subject has an average weekly alcohol intake of greater than 21 units if male or 14 units if female.
* The subject has any history of breathing problems (e.g. history of asthmatic symptoms).
* The subject is infected with the hepatitis B, hepatitis C, or HIV virus.
* The subject has had a respiratory tract infection or worsening of asthma within 4 weeks of the start of the study.
* The subject has a past or present disease, which as judged by the Investigator, may affect the outcome of this study.
* The subject has a history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxia seizures.
* The subject has taken inhaled, nasal or dermal steroids within 4 weeks or oral steroids within 8 weeks of the start of the study.
* The subject is unable to abstain from other drugs that may interfere with the conduct of the study.
* The subject has ongoing rhinitis that requires treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-02-07 (Actual); Primary Completion 2006-04-10 (Actual); Study Completion 2006-04-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability parameters will be compared between active and placebo treatment groups using summary statistics. No formal statistical analyses of the safety and tolerability data will be performed. | Up to 18 weeks

SECONDARY OUTCOMES:
Derived GW805858 and GW288967 PK parameters will be compared between active and placebo treatment groups using summary statistics. | Pre-dose, 5,20,30,45,60,90 minutes, 2,3,4,6,8,10,12,12.5,13,14, 24 hours Post-dose on Days 1 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study SF2105450 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/SF2105450?search=study&study_ids=SF2105450#rs